CLINICAL TRIAL: NCT00972803
Title: The Effects of Pistacia Mutica on De Novo Dental Plaque Formation, Gingival Inflammation and Oral Microorganisms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tabriz University (Other)
Responsible Party: Dr. Reza Pourabbas, Faculty of Dentistry, Tabriz Univ. of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8660
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2007-02

CONDITIONS: Gingivitis
Keywords: gingivitis; dental plaque; mouthrinse
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- pistacia Mutica (Experimental): The subjects were asked to use a mouthwash containing pistacia Mutica extract twice a day for 4 days.
  Interventions: Drug: pistacia Mutica extract
- placebo (Placebo Comparator): The subjects were asked to use a mouthwash containing Placebo twice a day for 4 days.
  Interventions: Drug: Placebo
- Chlorhexidine (Active Comparator): The subjects were asked to use a mouthwash containing Chlorhexidine twice a day for 4 days.
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: pistacia Mutica extract — The subjects were asked to use a mouthwash containing pistacia Mutica extract twice a day for 4 days.
  Arms: pistacia Mutica
Drug: Placebo — The subjects were asked to use a placebo mouthwash twice a day for 4 days.
  Arms: placebo
Drug: Chlorhexidine — The subjects were asked to use a mouthwash containing Chlorhexidine twice a day for 4 days.
  Arms: Chlorhexidine

SUMMARY:
Dental plaque is a well known etiologic factor for gingivitis. Recently, herbal extracts are a matter of scientific interest to inhibit plaque accumulation on teeth. The purpose of this study was to evaluate the effects of pistacia Mutica (PM) mouth wash on de novo dental plaque plaque formation, gingival inflammation indices and oral microorganisms.

ELIGIBILITY:
Inclusion Criteria:

* had merely gingivitis (pocket depth≤3 mm, no attachment loss)
* without any fixed or removable oral appliances

Exclusion Criteria:

* Individuals who had a history of any relevant systemic diseases
* Individuals who had a history of any drug usage

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The effects of pistacia Mutica extract (PM) on de novo plaque formation. | In a 4 days experimental periods followed by a 10 days wash-out periods.

SECONDARY OUTCOMES:
staining effects of pistacia Mutica extract in comparison to placebo or Chlorhexidine | In a 4 days experimental periods followed by a 10 days wash-out periods

CONTACTS AND LOCATIONS:
Overall Officials: Reza Pourabbas, DDS,MSD, Principal Investigator — Tabriz University of Medical Sciences
Locations (1):
- Drug Applied Science Center, tabriz Univ. of Medical Sciences, Tabriz, East Azerbaijan Province, Iran